CLINICAL TRIAL: NCT07020637
Title: Assessment of Stroke Volume in Shock Using Echocardiography Versus Bioreactive Impedance
Status: Recruiting | Type: Observational
Sponsor: University of Nevada, Las Vegas (Other)
Responsible Party: Sponsor
Other Study IDs: UNLV-2024-124
Record Dates: First submitted 2025-06-05; First posted 2025-06-13 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2024-12

CONDITIONS: Shock; Critical Illness
Keywords: Cheeta NICOM; Bioreactance; Transthoracic Echocardiography; Passive Leg Raising; Stroke Volume; Shock Assssment; Noninvasive Cardiac Output Monitoring
MeSH Terms: conditions — Shock; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Shock Patients: This cohort includes adult patients presenting with clinical signs of shock in the intensive care unit. Each participant will undergo stroke volume measurement using both transthoracic echocardiography and bioreactance-based monitoring (Cheetah NICOM) before and after passive leg raising. No therapeutic intervention will be performed as part of the study.
  Interventions: Device: Cheetah NICOM

INTERVENTIONS:
Device: Cheetah NICOM — Bioreactance-based noninvasive cardiac output monitoring device used to measure stroke volume before and after passive leg raising. Used solely for observational measurement. No therapeutic intervention is performed.

SUMMARY:
This study aims to evaluate the correlation between stroke volume measurements obtained by transthoracic echocardiography and bioreactance-based noninvasive cardiac output monitoring. The primary objective is to assess the level of agreement between these two modalities in critically ill patients.

DETAILED DESCRIPTION:
In this prospective observational study, patients presenting with clinical signs of shock will be enrolled after obtaining informed consent. Stroke volume (SV) will be measured using both transthoracic echocardiography and bioreactance-based noninvasive cardiac output monitoring (Cheetah NICOM). SV will be recorded before and after passive leg raising (PLR) to evaluate the correlation between the two methods in terms of absolute values and directional changes (increase or decrease). No therapeutic intervention will be performed as part of the study; all clinical decisions will remain under the discretion of the treating medical team.

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 18 years
* Clinical diagnosis of shock as determined by the treating ICU physician (e.g., hypotension requiring vasopressors or evidence of end-organ hypoperfusion)
* Able to obtain informed consent from the patient or a legally authorized representative
* Enrollment within 24 hours of ICU admission

Exclusion Criteria:

* Pregnancy
* Known severe aortic valve disease or dynamic left ventricular outflow tract obstruction
* Morbid obesity (BMI > 40) that precludes accurate echocardiographic imaging Presence of cardiac arrhythmias (e.g., atrial fibrillation with rapid ventricular response) affecting stroke volume measurements
* Implanted cardiac assist devices (e.g., LVAD, pacemaker dependency)
* Imminent death or decision for comfort care only

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to the intensive care unit (ICU) with clinical signs of shock, including hypotension and/or evidence of end-organ hypoperfusion, who are able to provide informed consent or have a legally authorized representative available.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-10-19 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Correlation Between Stroke Volume Measurements by Echocardiography and Bioreactance Monitoring | Within 1 hour of enrollment
  Pearson correlation coefficient between stroke volume measurements obtained using transthoracic echocardiography and those obtained using bioreactance-based monitoring (Cheetah NICOM) in response to passive leg raising.

CONTACTS AND LOCATIONS:
Overall Officials: Mutsumi J Kioka, Medical Doctor, Principal Investigator — UNLV
Locations (1):
- University Medical Center Southern Nevada, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to privacy concerns and the limited scope of this single-center observational study. No long-term data storage or external data-sharing infrastructure has been established for this project.